CLINICAL TRIAL: NCT06318403
Title: Estradiol Supplementation and Rotator Cuff Repair: A Preliminary Randomized Trial
Brief Title: Estradiol Supplementation and Rotator Cuff Repair
Acronym: ESTRCR
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Peter Chalmers, Associate Professor of Orthopaedic Surgery, Principal Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 177012
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Rotator Cuff Tears; Rotator Cuff Injuries; Rotator Cuff Syndrome; Menopause Related Conditions; Menopause
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transdermal estradiol patches (Experimental): All patients will receive patches with identical labeling from our pharmacy, to be applied twice weekly. In the study group, these will contain 0.025 mg/day of estradiol. In the control group, these will be placebo. These will be applied twice weekly for three months beginning at the time of surgery and extending for three months after surgery.
  Interventions: Drug: Transdermal estrogen; Procedure: Rotator Cuff Repair Surgery
- Placebo patches (Placebo Comparator): All patients will receive patches with identical labeling from our pharmacy, to be applied twice weekly. In the study group, these will contain 0.025 mg/day of estradiol. In the control group, these will be placebo. These will be applied twice weekly for three months beginning at the time of surgery and extending for three months after surgery.
  Interventions: Procedure: Rotator Cuff Repair Surgery

INTERVENTIONS:
Drug: Transdermal estrogen — All patients will receive patches with identical labeling from our pharmacy, to be applied twice weekly. In the study group, these will contain 0.025 mg/day of estradiol. In the control group, these will be placebo. These will be applied twice weekly for three months beginning at the time of surgery and extending for three months after surgery.
  Arms: Transdermal estradiol patches
Procedure: Rotator Cuff Repair Surgery — The operative protocol will be standardized in all patients. Both the operative protocol and post-operative rehabilitation protocol will be per our standard of care, without alteration. An arthroscopic approach will be used. In all cases a double-row rotator cuff repair using triple-loaded anchor(s) on the medial row will be used. Post-operatively all patients will be placed in a sling for six weeks. Active range of motion exercises will begin at six weeks post-operatively and strengthening will be delayed until 12 weeks post-operatively. In all phases of care our peri-operative and post-operative protocol for study patients will be similar to our current clinical practice to ensure generalizability.

SUMMARY:
Rotator cuff tears in the shoulder are common causes of pain and disability, often fail to heal with surgery, and tears, worse outcomes after surgery, and failure of healing are associated with estradiol deficiency. In this study, post-menopausal women will be randomized to either estradiol patches or placebo patches after repair of the rotator cuff. The purpose of this study is to determine whether estradiol patches show promise in improving shoulder pain, strength, muscle volumes, and function when given with rotator cuff repair.

DETAILED DESCRIPTION:
Injuries to the rotator cuff are among the most common musculoskeletal complaints and are increasing in incidence. Multiple studies have demonstrated that rotator cuff repair (RCR) improves outcomes for rotator cuff tears. Over 500,000 RCRs are performed in the US annually. When both surgical and non-operative treatment are included, rotator cuff injuries cost the United States over $5 billion dollars annually. After RCR, tendon healing fails to occur in >20% of patients. Improving tendon healing is thus a critical barrier to success. The field has arrived at a consensus that improving tendon biology is the key to improving tendon healing. Our prior human and animal research demonstrates that estradiol deficiency contributes to rotator cuff injuries and poor outcomes after RCR and estradiol supplementation improves RCR healing and outcomes. With this study we propose to translate these promising and compelling findings into improved clinical care of patients with rotator cuff injuries. Estradiol deficiency can be treated with hormone therapy (HT), which is widely utilized, well-tolerated, inexpensive, and FDA approved. In this study, we will conduct a phase II study of the efficacy and feasibility of HT within the setting of RCR. We hypothesize that compliance and response rates will be high while adverse events will be infrequent and equally common with estradiol patches and placebo patches. We also hypothesize that outcomes and healing will be better in the HT group than the control group. To test these hypotheses, we will conduct a randomized, placebo-controlled, double-blinded clinical trial to measure recruitment and retention rates, compliance with treatment, response to treatment of serum hormone levels, estimated effect size for power calculations, and adverse events. Postoperatively, we will evaluate validated patient-reported outcomes and tendon healing and rotator cuff muscle volumes utilizing magnetic resonance imaging. If efficacy and tolerability are demonstrated, a future large, multi-center, randomized clinical trial will be warranted. We expect these data will support the use of estradiol as a promising approach to improved healing and outcomes, supporting a future, larger, well-powered, multi-centered randomized clinical trial with longer follow-up. Such a study could improve the treatment of people with rotator cuff injuries, thereby decreasing a source of significant disability. If our hypotheses are confirmed, it would shift the paradigm on the treatment of problems with tendons and their attachments to bone throughout the body.

ELIGIBILITY:
Inclusion Criteria

1. A plan for a primary rotator cuff repair
2. Female sex (assigned sex at birth)
3. >1 cm tear width, full thickness supraspinatus/infraspinatus tear
4. Post-menopausal, as defined by at least twelve months since last menses
5. Age 50-80

Exclusion Criteria

1. Active infection
2. Baseline serum estradiol >20 pg/mL
3. Infraspinatus or supraspinatus muscle atrophy of greater than or equal to Goutallier grade 3
4. Pre-operative systemic estradiol supplementation
5. Medically unfit for operative intervention
6. Revision surgery
7. Unwillingness to participate in the study, including post-operative imaging
8. Inability to read or comprehend written instructions
9. Prisoner
10. Concomitant patch augmentation or tendon-transfer
11. Breast cancer or a history of breast cancer or other estradiol-dependent neoplasia
12. Liver disease as documented in the medical record
13. Active venous thromboembolic disease, such as deep venous thrombosis, pulmonary embolism, a history of these conditions, or a known predisposition to these disorders (such as Protein C, protein S, or antithrombin deficiency)
14. Active arterial thromboembolic disease, such as stroke, myocardiac infarction, a history of these conditions, or a known predisposition to these disorders
15. Isolated subscapularis tears
16. Known anaphylactic reaction or hypersensitivity to estradiol, adhesive, or transdermal patches

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
American Shoulder and Elbow Surgeons (ASES) Score | To be collected within 3 months pre-operatively and at 6 weeks (±2 weeks), 12 weeks (±2 weeks), and 6 months (±4 weeks) post-operatively.
  The ASES score is a patient survey that creates a score on a 100 point scale incorporating questions regarding shoulder pain and shoulder function. This survey contains 11 questions and takes ~3 minutes to complete. The validity and reliability of this score has been previously validated.

SECONDARY OUTCOMES:
Simple Shoulder Test (SST) Score | To be collected within 3 months pre-operatively and at 6 weeks (±2 weeks), 12 weeks (±2 weeks), and 6 months (±4 weeks) post-operatively.
  The SST score is a patient survey that creates a score on a 12-point scale incorporating questions regarding shoulder function. This survey contains 12 questions and takes ~3 minutes to complete. The validity and reliability of this score has been previously validated.
Visual Analogue Score (VAS) for pain | To be collected within 3 months pre-operatively and at 6 weeks (±2 weeks), 12 weeks (±2 weeks), and 6 months (±4 weeks) post-operatively.
  The VAS pain score is a patient survey that creates a score on a 10 point scale incorporating a single question regarding shoulder pain. This survey takes <1 minute to complete.
Magnetic Resonance Imaging (MRI) | Within 3 months pre-operatively and at 6 months (±4 weeks) post-operatively.
  MRI scans will be assessed by observers blinded to the patient's allocation. On the pre-operative MRI, pre-operative tear width, pre-operative tear retraction, cuff muscle atrophy using the Goutallier10 classification will be measured. For each patient, the post-operative MRI will be classified using the Sugaya classification, which multiple authors have demonstrated to have excellent inter-observer reliability. Sugaya grades 1, 2, and 3 will be considered "healed" and Sugaya grades 4 and 4 will be considered "re-torn". In cases of re-tear, tear width and retraction will be measured. In addition, on both pre-operative and post-operative scans rotator cuff muscle volumes will be measured, for which we have previously demonstrated to have excellent inter-observer reliability and accuracy. All post-operative MRI scans will be 3.0 tesla non-arthrogram studies in which T2 imaging will be performed in the sagittal, coronal, and axial planes.
Strength Assessment | To be collected within 3 months pre-operatively and at 6 weeks (±2 weeks), 12 weeks (±2 weeks), and 6 months (±4 weeks) post-operatively.
  Rotator cuff strength, as measured with a handheld digital dynamometer (Lafayette instruments, Lafayette, IN), will be measured. Abduction strength will be measured at 30 degrees of flexion, 30 degrees of abduction, neutral rotation, and full elbow extension. External rotation strength will be measured with the arm in adduction, neutral rotation, and 90 degrees of elbow flexion. These measures will be performed by research coordinators trained to perform these assessments. We have previously demonstrated these measurements to have excellent inter-observer reliability, with abduction strength having an intra-class correlation coefficient (ICC) of 0.993 and external rotation strength having an ICC of 0.986.
Range of motion | To be collected within 3 months pre-operatively and at 6 weeks (±2 weeks), 12 weeks (±2 weeks), and 6 months (±4 weeks) post-operatively.
  Range of motion will be recorded. Research personnel experienced with the use of video will measure active abduction, active forward elevation, active internal rotation in adduction, and active external rotation in adduction. This protocol has been previously used in many publications. These videos will be saved using subject numbers and then evaluated using a digital protractor by a third-party observer blinded to the subjects group. This method of range of motion measurement has been previously demonstrated to have excellent inter-observer reliability.

OTHER OUTCOMES:
Serum Hormone Measurement | To be collected within 3 months pre-operatively, at 6 weeks (±1 week) after starting medication, and at 12 weeks (±2 weeks) after starting medication.
  Nonadherence could result in cross-over, biasing towards the null hypothesis. We will assess compliance with serum laboratory values. Blood will be drawn and the following serum estradiol values will be collected. These values will be interpreted by co-investigator Dr. Corrine Welt, a board-certified endocrinologist with extensive experience with reproductive urology. To preserve participant blinding, the results of hormonal testing will not be available through the patient electronic portal unless it is deemed necessary for patient care by Dr. Welt. In addition, to preserve their blinding, the treating surgeons and the clinical research coordinators performing the post-operative assessments will not have access to the laboratory values. Dr. Welt will not perform any other patient evaluations, and thus cannot influence the results.
Patch Count | 6 weeks (±2 weeks) post-operatively, 12 weeks (±2 week) post-operatively.
  Subjects will be asked how many patches they have used to determine patient compliance. Deviations from protocol will be recorded.
Averse Event Assessment | To be collected at every patient visit, including 6 weeks (±2 weeks) after surgery, 12 weeks (±2 weeks) after surgery, and 6 months (±4 weeks) after surgery.
  At each visit patients will be queried regarding adverse events. Patients will asked about the following specific adverse events side effects: dyspepsia/gastritis, hypertension, flu-like symptoms, back-pain, headache, anxiety, insomnia, depression, breast tenderness, vaginal bleeding, hot flashes, venous insufficiency, vertigo, edema, deep venous thrombosis, application site reactions, abdominal pain, weight gain, emotional lability, bleeding, infection, complications from anesthesia, the need for further surgery. In addition, any post-operative injections will be recorded.

IPD SHARING:
Plan to Share IPD: No
The authors will plan to make their results available through multiple venues. Our plan includes the following:
  1. Presentation at national scientific meetings.
  2. ClinicalTrials.gov.
  3. Publication in peer-reviewed literature.
  4. Data sharing upon request. The PI will provide de-identified data to those who make requests for the purposes of meta-analysis.
  5. Visiting Professors.
  6. Website. The University of Utah regularly publishes important research results in web log ("blog") format, as does the PI on his practice website. Summaries of these results, along with links to the full results, written primarily for a general audience, will be posted as they become available.
  7. Repository. Once the main findings are accepted for publication, the final dataset will be shared at https://dataverse.org. This will be performed after removal of all protected health information.
  8. Progress on data sharing will be reported in our Research Progress Performance Reports annually.